CLINICAL TRIAL: NCT03615222
Title: The Impact of Modifiable Psychosocial Factors on Veterans' Long-term Trajectories of Functioning and Quality of Life: Promoting Recovery by Targeting Mindfulness and Psychological Flexibility
Brief Title: Impact of Modifiable Psychosocial Factors on Veterans' Long-term Trajectories of Functioning and Quality of Life
Acronym: SERVE:IMPACT
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D0304-I
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: PTSD; Depression; Chronic Pain; Alcohol Use Disorder; Traumatic Brain Injury
Keywords: functional impairment; quality of life; Veterans; mindfulness; Acceptance and Commitment Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Chronic Pain; Alcoholism; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva optionally collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SERVE assessment only: Eligible veterans will complete 4 assessments over a two year period of time.

SUMMARY:
This study is Phase 3 of Project SERVE (Study Evaluating Returning Veterans' Experiences). Through two prior phases, SERVE has followed a cohort of post-9/11 Veterans since 2010 and has identified numerous risk and protective factors. SERVE's overall objective is to understand and improve the long-term functional outcomes of post-9/11 Veterans. Consistent with the investigators' conceptual model, the central hypothesis is that psychological flexibility and other trans-diagnostic treatment targets mediate the effects of the most common mental and physical wounds of war on long-term functioning and self-directed violence (i.e., suicide risk). Thus, integrated interventions specifically designed to improve functioning associated with these conditions are most likely to promote long-term recovery among the most impaired Veterans. The investigators will test the central hypothesis and accomplish the overall objective by pursuing the following specific aims:

Aim 1: Identify treatment targets that prospectively predict functional disability, family functioning and self-directed violence (SDV) in post-9/11 Veterans with PTSD, depression, chronic pain, TBI, and/or AUD.

To achieve this aim, the investigators will follow 500 Veterans for 2 years in order to prospectively evaluate the impact of several novel, treatment-relevant factors on functional disability and SDV over time.

H1: Novel factors (mindfulness, perceived burdensomeness, thwarted belongingness, and moral injury) along with established treatment targets (psychological flexibility, self-compassion, and emotion regulation) will prospectively predict functional disability and SDV after accounting for covariates.

DETAILED DESCRIPTION:
Research by the investigators' team and others demonstrates that posttraumatic stress disorder (PTSD), depression, alcohol use disorders (AUD), traumatic brain injury (TBI), and chronic pain frequently co-occur among post-9/11 war Veterans and are associated with functional impairment and suicide risk; however, no treatment currently exists that has been specifically designed to promote functional recovery among Veterans experiencing any combination of these most common mental and physical wounds of war. The investigative team has: (A) identified multiple modifiable psychosocial factors (emotion regulation, psychological flexibility, self-compassion) that prospectively predict impairment and suicidal ideation in Veterans; (B) characterized long-term trajectories of resilience and functional disability in Veterans; (C) determined that high utilization of VA mental health services appears to have little, if any, impact on the functional recovery of Veterans on the moderate and severely impaired trajectories; (D) identified psychological flexibility (i.e., the ability to remain present in the moment despite emotional distress and to persist in changing behavior in the pursuit of one's values and goals) as a unique, prospective predictor of membership in the severely impaired functional trajectory and of suicidal ideation, even after accounting for the effects of co-morbidity; and (E) demonstrated that Acceptance and Commitment Therapy (ACT)-a trans-diagnostic, mindfulness-based behavior therapy that seeks to improve functioning by targeting psychological flexibility -can lead to recovery, including sustained improvements in functional disability, quality of life (QoL), suicidal ideation, PTSD, and AUD symptoms among severely impaired Veterans with co-occurring PTSD-AUD.

This study is Phase 3 of Project SERVE (Study Evaluating Returning Veterans' Experiences). Through two prior RR&D MERIT awards, SERVE has followed a cohort of post-9/11 Veterans since 2010 and has identified numerous risk and protective factors. SERVE's overall objective is to understand and improve the long-term functional outcomes of post-9/11 Veterans. Consistent with the investigators' conceptual model, the central hypothesis is that psychological flexibility and other trans-diagnostic treatment targets mediate the effects of the most common mental and physical wounds of war on long-term functioning and self-directed violence (i.e., suicide risk). Thus, integrated interventions specifically designed to improve functioning associated with these conditions are most likely to promote long-term recovery among the most impaired Veterans. The investigators will test the central hypothesis and accomplish the overall objective by pursuing the following specific aims:

Aim 1: Identify treatment targets that prospectively predict functional disability, family functioning and self-directed violence (SDV) in post-9/11 Veterans with PTSD, depression, chronic pain, TBI, and/or AUD.

To achieve this aim, the investigators will follow 500 Veterans for 2 years in order to prospectively evaluate the impact of several novel, treatment-relevant factors on functional disability and SDV over time.

H1: Novel factors (mindfulness, perceived burdensomeness, thwarted belongingness, and moral injury) along with established treatment targets (psychological flexibility, self-compassion, and emotion regulation) will prospectively predict functional disability and SDV after accounting for covariates.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the longitudinal assessment study are as follows:

* Potential participants include male and female
* English-speaking OEF/OIF/OND Veterans
* Enrolled at CTVHCS or willing to be enrolled for the purpose of participation in this study.

To be eligible, participants must be

* able to comprehend and sign the informed consent form
* able to complete the structured interviews and self-report assessments
* willing to be contacted for follow-up assessments

For newly enrolled participants:

* given that the investigators have already recruited a large sample of veterans who are reporting relatively little functional impairment, the investigators will require newly enrolled participants to self-report global functional impairment on the WHODAS 2.0 12-item self-report version equivalent to a mean item score of 1.0.

  * Although the investigators anticipate being able to meet the recruitment goals, should recruitment prove more challenging than expected, the investigators will remove this inclusion criterion
* deemed stable on psychotropic medications (defined as 3 months on a selective serotonin reuptake inhibitor or monoamine oxidase inhibitor; >1 month on an anxiolytic or beta-blocker; >1 month medication discontinuation or "wash out" for all medications) at the time of the BL assessment
* deemed stable in psychotherapy (3 months stabilization for psychotherapy and 1-month psychotherapy wash-out) at the time of the BL assessment

  * These latter two criteria are instated to ensure that symptoms assessed during the baseline assessment are due to any underlying psychiatric condition and not due to the effects of starting or stopping medications and/or psychotherapy.
* Changes in treatment will be permissible during the current study, as this reflects real-world practice
* All changes in medications will be monitored over time, and appropriately covaried, as treatment can have important effects on functioning over time
* Individuals will be eligible to participate with current and lifetime psychiatric diagnoses, with the exception of:

  * schizophrenia
  * schizophreniform disorder
  * schizoaffective disorder
  * delusional disorder
  * unspecified schizophrenia spectrum/other psychotic disorder, and bipolar disorder

Additional inclusion criteria specific to the SCD treatment study are:

* Veterans will have a global disability (mean item) score on the WHODAS 2.0 of 1.0, which is 1 SD above the mean of the large non-psychiatric sample of Veterans from SERVE and VA Boston during both of their last 2 assessments

Exclusion Criteria:

Exclusion criteria for the longitudinal assessment study are as follows:

* plan to relocate out of the CTVHCS system within four months of protocol initiation
* meet criteria for a diagnosis of:

  * schizophrenia
  * schizophreniform disorder
  * schizoaffective disorder
  * delusional disorder
  * a manic/hypomanic episode
* report current suicidal or homicidal risk warranting crisis intervention
* report symptoms consistent with severe traumatic brain injury (TBI) that interfere with their ability to complete the consent process or assessment

  * i.e., due to ethical concerns about obtaining informed consent and difficulties with completing the structured assessment
* report current non-military related hallucinations or delusions that cause significant distress and/or impairment

Additional exclusion criteria for the SCD treatment study are:

* recent (1 month) or anticipated change in psycho-pharmacological treatment. Veterans may stay on current medications but will be asked to refrain from changes to the extent possible based on safety
* logistical circumstances that would interfere with study completion
* Presence of a non-alcohol substance use disorder (SUD) deemed to be the primary focus of treatment

  * Those with a principal AUD will be eligible.
* Additional diagnoses of non-alcohol SUD are allowed, unless they are deemed the principal focus of treatment.
* Potentially eligible Veterans who score above the clinical cutoff on the DAST will be asked additional questions during the eligibility screening to determine whether they meet criteria for a principal non-alcohol SUD (see phone screen)
* AUD/SUD of sufficient severity that residential, rather than outpatient, treatment is indicated based on potential safety concerns associated with withdrawal.

  * This determination will be made by the PI, with consultation from the Veteran's existing treatment providers, as appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzannah K. Creech, PhD, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (2):
- United States (2):
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Upon written request by qualified researchers and following institutional guidelines, deidentified data may be shared if the study participant consented to data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within one year of completion of the study
Access Criteria: Upon written request by qualified researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SERVE Assessment Only
Started | 377
Completed | 343
Not Completed | 34
Not completed — Ineligible | 26
Not completed — Withdrawal by Subject | 7
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Analyses include only eligible participants (n=351).
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 340
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.20 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60
  Not Hispanic or Latino | 291
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 103
  White | 187
  More than one race | 32
  Unknown or Not Reported | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 351
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Self-report of symptoms of PTSD during the previous month. Demonstrates high sensitivity and specificity in relation to a lengthy diagnostic interview for PTSD (CAPS), with which it was co-developed. Total scores range from 0 to 80 with higher scores indicating more symptoms of PTSD. Provisional PTSD diagnosis 33+.
  units on a scale | 27.47 (20.77)
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Self-report measure to screen for alcohol-use disorders (Saunders, Aasland, Babor, Fuente, & Grant, 1993). 10-item measure adopted by VA as the gold-standard screening for alcohol use disorders in mental health and primary care clinics. Good internal consistency (α=.80-.94) and test-retest reliability (r=.86), and strong concurrent validity with the MAST and CAGE screening measures (Babor et al., 2001). Total scores range from 0 to 40 with higher scores indicating more problematic drinking behavior. Non-drinker (0); Hazardous/Harmful Alcohol Consumption (8-14); Provisional AUD diagnosis (15+).
  units on a scale | 3.54 (5.12)
Drug Abuse Screening Test (DAST-10) [Mean (Standard Deviation); unit: units on a scale] — Self-report measure to quantify drug misuse and related psychosocial impairment. Good internal consistency and concurrent validity with frequency of drug use over 12-months (Skinner, 1982). Moderately correlated with denial and social desirability. The instructions will be updated to more explicitly assess for misuse of opiates that may have been prescribed. Total scores range from 0 to 10 with higher scores indicating more problems with drug use. No problems (0); Low level (1-2); Moderate level (3-5); Substantial level (6-8); Severe level (9-10).
  units on a scale | 1.13 (.97)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Self-report measure used for screening, diagnosing, and monitoring depression. It incorporates DSM-V diagnostic criteria (Question 9 screens for suicidal ideation; Kroenke, Spitzer & Williams, 2001). Total scores range from 0 to 27 with higher scores indicating more symptoms of depression. Mild (5-9); Moderate (10-14); Moderately Severe (15-19); Severe (20-27).
  units on a scale | 10.09 (6.56)

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Scale
Description: The Columbia Suicide Severity Rating Scale (C-SSRS; Posner et al., 2008) is a state-of-the-art suicide assessment for individuals perceived to be at high risk for suicidality. Internal consistency ranged from .73 to .95 (Posner et al., 2011). Values on the intensity of suicidal ideation (e.g., frequency, duration, controllability, deterrents, reasons for ideation) are summed to create a total score; range from 0 to 25, where higher scores indicate higher SI severity.
Time Frame: Baseline and 24-month
Population: Analysis at 24-month includes the 216 participants who completed the clinical assessment at follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
score on a scale
  Baseline | 1.19 (3.76)
  24-month: number analyzed (Participants) | 216
  24-month | 1.09 (3.67)

2. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: Self-report assessment of functional disability with total score and 6 domains of functioning: understanding and communicating, mobility, getting along with others, life activities (i.e., work, education, household responsibilities), participation in society, and self-care (Ustun et al., 2010). Both global and specific areas of functioning are crucial in thoroughly understanding functional recovery, as Veterans may function well in one area and have difficulty in another. Moreover, some domains may be affected by contextual factors instead of representing functional capacity (e.g., work functioning in a struggling economy independent of impairment). Means on this measure capture items from all domain subscales and can range from 0 to 3 where higher scores indicate higher levels of disability.
Time Frame: Baseline, 8-month, 16-month, and 24-month
Population: Differences in participants reflect number completed at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
score on a scale
  Baseline | 1.20 (.80)
  8-month: number analyzed (Participants) | 319
  8-month | 1.28 (.77)
  16-month: number analyzed (Participants) | 306
  16-month | 1.21 (.80)
  24-month: number analyzed (Participants) | 297
  24-month | 1.03 (.79)

3. Primary Outcome: Clinician Administered NSSI Disorder Index (CANDI)
Description: The Clinician Administered NSSI Disorder Index (CANDI) is a clinical interview that diagnoses Nonsuicidal Self Injury (NSSI) disorder and type and frequency of NSSI. Demonstrated good reliability and validity in prior research. Results report the number of participants that meet for a diagnosis of NSSID.
Time Frame: Baseline and 24-month
Measure: Count of Participants; unit: Participants
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
Participants
  Baseline - Lifetime NSSID | 31
  Baseline - Current NSSID | 8
  24-month - Current NSSID | 5

4. Primary Outcome: Inventory of Psychosocial Functioning (IPF) - Brief
Description: Self-report measure (Marx et al., 2009; Bovin et al., 2018) of problems in different domains of life (e.g., Romantic Relationships with a Spouse/Partner, Family, Work, Friendships and Socializing, Parenting, Education, and Self-Care). The short version has a .90 correlation with the full 80-item instrument (Co-I Marx, personal communication). Adjusted totals range from 0 to 100 with higher scores indicate greater functional impairment.
Time Frame: Baseline, 8-month, 16-month, and 24-month
Population: Differences in participants reflect number completed at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
score on a scale
  Baseline | 44.96 (23.06)
  8-month: number analyzed (Participants) | 318
  8-month | 48.02 (22.64)
  16-month: number analyzed (Participants) | 305
  16-month | 46.04 (22.85)
  24-month: number analyzed (Participants) | 297
  24-month | 39.89 (23.46)

5. Primary Outcome: Beck Scale for Suicide Ideation (BSSI)
Description: Widely-used self-report measure of intensity of thoughts and behaviors associated with suicide. Includes 2 additional items that ask about past suicide attempts as well as the level of suicidal intent during the most recent attempt. Prior research shows that endorsement of suicidal thoughts and behaviors can be greater on self-report questionnaires compared to interviews. Total scores range from 0 to 42 where higher scores indicate higher suicidal ideation.
Time Frame: Baseline and 24-month
Population: Differences in participants reflect number completed at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
score on a scale
  Baseline | 1.99 (4.66)
  24-month: number analyzed (Participants) | 292
  24-month | 1.61 (4.16)

6. Primary Outcome: Quality of Life Scale
Description: Self-report (Burkhardt, et al., 1989) assessing how satisfied people are in different areas of their life, distinct from health status, (e.g., mate, physical well-being, relationships with others, social, community, and civic activities, personal development and fulfillment, recreation, and independence). Good internal consistency and high test-retest reliability (Burckhardt et al. 2003). Total scores range from 16 to 112 with higher scores indicating greater life satisfaction.
Time Frame: Baseline, 8-month, 16-month, and 24-month
Population: Differences in participants reflect number completed at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SERVE Assessment Only
Number analyzed (Participants) | 351
score on a scale
  Baseline | 75.03 (18.39)
  8-month: number analyzed (Participants) | 319
  8-month | 72.09 (18.35)
  16-month: number analyzed (Participants) | 306
  16-month | 73.38 (18.90)
  24-month: number analyzed (Participants) | 292
  24-month | 76.56 (19.18)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | SERVE Assessment Only
All-Cause Mortality (participants affected / at risk) | 1/351
Serious Adverse Events (participants affected / at risk) | 25/351
Other Adverse Events (participants affected / at risk) | 0/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SERVE Assessment Only (N=351)
Mental Health Hospitalization (Psychiatric disorders) | 5 (5) — Hospitalized following an increase of mental health symptoms and/or suicide attempt
Jailed (General disorders) | 4 (4) — Reported being jailed overnight
Minor Surgery (General disorders) | 16 (16) — Overnight hospitalization for minor surgery

LIMITATIONS AND CAVEATS:
Due to COVID-19 there was a pause in data collection which lead to fewer participants than originally targeted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03615222/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03615222/ICF_001.pdf